CLINICAL TRIAL: NCT04192149
Title: The Effects of Ultrasound on Central Nervous System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 21331
Record Dates: First submitted 2019-03-19; First posted 2019-12-10 (Actual); Last update posted 2019-12-10 (Actual); Status verified 2019-12

CONDITIONS: Focused Ultrasound
Keywords: Ultrasound; Neuromodulation; Focused Ultrasound

STUDY DESIGN:
Intervention Model Description: Within subjects design of focused ultrasound and control
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Patients receiving Craniotomy (Experimental): Patients receiving an awake or asleep craniotomy for brain tumors and/or epilepsy will undergo a brain mapping procedure using electrical stimulation as a part of their normal care. The research procedures will duplicate this mapping with an invasive Focused Ultrasound mapping.
  Interventions: Other: Focused Ultrasound
- Epilepsy Patients (Experimental): Patients undergoing long term monitoring for epilepsy will receive a non-invasive form of Focused Ultrasound stimulation which will be measured by their EEG cap and intracranial electrodes which are a part of their normal care.
  Interventions: Other: Focused Ultrasound
- Tremor Patients receiving FUS (Experimental): Patients undergoing high intensity FUS treatment for tremor will be asked to wear a research provided EEG cap while undergoing a non-invasive low intensity Focused Ultrasound research procedure and changes in their tremor will be monitored.
  Interventions: Other: Focused Ultrasound
- Tremor Patients receiving DBS (Experimental): Patients undergoing Deep Brain Stimulation (DBS) treatment for tremor will receive a non-invasive Focused Ultrasound stimulation observed through their newly implanted electrode.
  Interventions: Other: Focused Ultrasound
- Patients receiving Spinal Surgery (Experimental): Patients receiving a spinal surgery will undergo a spinal stimulation using electrical stimulation as a part of their normal care. The research procedures will duplicate this with an invasive Focused Ultrasound stimulation.
  Interventions: Other: Focused Ultrasound

INTERVENTIONS:
Other: Focused Ultrasound — Low intensity focused ultrasound is sound energy stimulation at a low intensity of 1-30 W/cm2

SUMMARY:
Focused ultrasound at low intensities is a form of neuromodulation with high spatial resolution that can be applied invasively or non-invasively using acoustic energy to affect neuronal activity. The purpose of this study is to better understand the effects of low intensity focused ultrasound (FUS) on the central nervous system. Specific patient populations within UVA health system are undergoing treatment that provide unique opportunities to study these effects.

DETAILED DESCRIPTION:
Focused ultrasound (FUS) at low intensities is a form of neuromodulation with high spatial resolution that can be applied invasively or non-invasively using acoustic energy to affect neuronal activity. In this study the investigators intended to use specific patient populations to investigate the effects of FUS on different areas of the central nervous system (CNS). Each of our patients groups is undergoing a unique procedure at University of Virginia that will provide us different insights into the CNS. (1) Patients receiving an awake or asleep craniotomy for brain tumors and/or epilepsy will undergo a brain mapping procedure using electrical stimulation as a part of their normal care. The research procedures will duplicate this mapping with an invasive FUS mapping. (2) Patients undergoing long term monitoring for epilepsy will receive a non-invasive form of FUS stimulation which will be measured by their EEG cap and intracranial electrodes which are a part of their normal care. (3) Patients undergoing high intensity FUS treatment for tremor will be asked to wear a research provided EEG cap while undergoing a non-invasive low intensity FUS research procedure and changes in their tremor will be monitored. (4) Patients undergoing Deep Brain Stimulation (DBS) treatment for tremor will receive a non-invasive FUS stimulation observed through their newly implanted electrode. (5) Patients receiving a spinal surgery will undergo a spinal stimulation using electrical stimulation as a part of their normal care. The research procedures will duplicate this with an invasive FUS stimulation.

ELIGIBILITY:
Inclusion Criteria:

* Be a patient receiving a treatment or surgical procedure specified below:
* Receiving a Craniotomy with brain mapping
* Receiving treatment or monitoring for Epilepsy
* Receiving either FUS or DBS treatment for Tremor
* Receiving a Spinal Surgery for stimulator placement
* Able to provide informed consent
* Must speak English
* Age 18-85

Exclusion Criteria:

* Not receiving one of the specified inclusion procedures
* Unable to provide consent
* Women who self-report pregnancy
* Patients who are currently incarcerated

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-02-19 (Actual); Primary Completion 2021-02-20 (Estimated); Study Completion 2021-02-20 (Estimated)

PRIMARY OUTCOMES:
Electrophysiological Changes as a result of Ultrasound | baseline, immediately after ultrasound (same day, approximately 5-10 minutes after baseline)
  Each participant group has different type of electrophysiological recording depending on the type of procedure. Recordings will include a baseline, during ultrasound, and/or post-ultrasound electrophysiology.

CONTACTS AND LOCATIONS:
Overall Officials: Wynn Legon, PhD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided